CLINICAL TRIAL: NCT06060626
Title: Optimization of Sedation Protocol for Endoscopic Procedures Using Impedance Ventilation Monitor.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ExSpironUVN
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2023-09

CONDITIONS: Sedation Complication; Ventilatory Depression
Keywords: sedation protocol; endoscopic procedure; ventilation monitoring; ventilatory depression
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Propofol; Fentanyl

STUDY DESIGN:
Intervention Model Description: The study will be performed on a sample of patients undergoing an endoscopic procedure requiring sedation. Patients will be divided into two groups, one group will be sedated with propofol only, the other will be premedicated with the opioid analgesic fentanyl before the procedure.
Who Masked: Care Provider
Masking Description: The endoscopist performing the procedure will not be informed which group the patient belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Active Comparator): Patients in whom only propofol will be administered during sedation. Intermittent boluses of propofol titrated to moderate level of sedation.
  Interventions: Drug: Sedation using only Propofol.
- Fentanyl (Active Comparator): Patients in whom combination of propofol and fentanyl will be administered during sedation.
  Fentanyl 1 ug/kg bolus 3 minutes before induction + Propofol intermittent boluses titrated to moderate level of sedation.
  Interventions: Drug: Sedation using combination of Propofol and Fentanyl.

INTERVENTIONS:
Drug: Sedation using only Propofol. — Patients in whom only propofol will be administered during sedation.
  Other Names: Propofol
  Arms: Propofol
Drug: Sedation using combination of Propofol and Fentanyl. — Patients in whom combination of propofol and fentanyl will be administered during sedation.
  Other Names: Fentanyl
  Arms: Fentanyl

SUMMARY:
The aim of the study is to evaluate the effect of opioids administered during sedation on patients' respiratory activity (ventilation) and comfort of the operator and patient during the endoscopic procedure. A common side effect of sedation is the effect on patients' ventilation, resulting from a combination of attenuation of respiratory centre activity and loss of patent airways. Shallow sedation will reduce these risks, but in addition to patient discomfort, it also increases the difficulty or impossibility of the endoscopist to perform the procedure. Choosing the appropriate method of sedation thus fundamentally affects the course of the procedure from the point of view of both the patient and the endoscopist. The aim is to prove that sedation with propofol alone compared to sedation with propofol and fentanyl premedication leads to the need for higher cumulative doses of administered propofol, higher risk of respiratory depression and lower patient and operator comfort. In addition, the non-invasive respiratory volume monitor (ExSpiron 2Xi) will be used for standard patient monitoring during the procedure, which assesses the lung tidal volume and respiratory rate by measuring the electrical impedance of the chest. This measurement captures inadequate ventilation before saturation drops, allowing even slight differences between selected drugs to be compared.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of opioids administered during sedation on patients' respiratory activity (ventilation) and comfort of the operator and patient during the endoscopic procedure. A common side effect of sedation is the effect on patients' ventilation, resulting from a combination of attenuation of respiratory centre activity and loss of patent airways. Shallow sedation will reduce these risks, but in addition to patient discomfort, it also increases the difficulty or impossibility of the endoscopist to perform the procedure. Choosing the appropriate method of sedation thus fundamentally affects the course of the procedure from the point of view of both the patient and the endoscopist. The aim is to prove that sedation with propofol alone compared to sedation with propofol and fentanyl premedication leads to the need for higher cumulative doses of administered propofol, higher risk of respiratory depression and lower patient and operator comfort. Standard monitoring during endoscopic procedures using sedation includes continual recording of ECG and respiratory rate (using the same electrodes), measurement of arterial blood oxygen saturation using a pulse oximeter and blood pressure measurement. Extended monitoring of spontaneous ventilation during sedation includes analysis of the concentration of exhaled carbon dioxide or analysis of the arterial blood gases.However, these methods have limitations and often critically reduced respiratory activity is diagnosed too late. Impedance monitoring of ventilation is now being introduced into clinical practice. In addition, the non-invasive respiratory volume monitor (ExSpiron 2Xi) will be used for standard patient monitoring during the procedure, which assesses the lung tidal volume and respiratory rate by measuring the electrical impedance of the chest. This measurement captures inadequate ventilation before saturation drops, allowing even slight differences between selected drugs to be compared.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled therapeutic or diagnostic colonoscopy with sedation
* Supine or lateral decubitus position
* Age 18-65
* American Society of Anesthesiologists (ASA) physical status classification system 1-2
* Informed consent signed

Exclusion Criteria:

* Planned frequent use of electrocoagulation
* Contact allergy for adhesive pads, excessive thoracic hair or other problem with pads
* contraindication of using Propofol or Fentanyl
* Incapability to understand the informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Incidence of significant decrease in ventilation during propofol sedation. | during the endoscopic procedure
  Incidence of significant decrease in ventilation during sedation with propofol alone during endoscopic surgery.
Incidence of significant decrease in ventilation during propofol and fentanyl sedation. | during the endoscopic procedure
  Incidence of significant decrease in ventilation during sedation with propofol and fentanyl during endoscopic surgery.

SECONDARY OUTCOMES:
Subjective assessment of the comfort of the procedure by the endoscopist. | immediately after the procedure
  Subjective assessment of the comfort of the procedure by the endoscopist using a questionnaire.
Subjective assessment of the comfort of the procedure by the patient. | immediately after the procedure
  Subjective assessment of the comfort of the procedure by the patient using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Trtíková, Mgr., Ph.D., Study Chair — CHARLES UNIVERSITY, FIRST FACULTY OF MEDICINE AND MILITARY UNIVERSITY HOSPITAL PRAGUE; David Novotný, M.D., Principal Investigator — CHARLES UNIVERSITY, FIRST FACULTY OF MEDICINE AND MILITARY UNIVERSITY HOSPITAL PRAGUE; Tomáš Tyll, M.D., Ph.D., Principal Investigator — CHARLES UNIVERSITY, FIRST FACULTY OF MEDICINE AND MILITARY UNIVERSITY HOSPITAL PRAGUE; Michal Soták, M.D., Ph.D., Principal Investigator — CHARLES UNIVERSITY, FIRST FACULTY OF MEDICINE AND MILITARY UNIVERSITY HOSPITAL PRAGUE
Locations (1):
- Military University Hospital Prague, Prague, Czechia, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Kassem MA, Zhou Y, Shabsigh M, Wang Q, Xu X. A Brief Review of Non-invasive Monitoring of Respiratory Condition for Extubated Patients with or at Risk for Obstructive Sleep Apnea after Surgery. Front Med (Lausanne). 2017 Mar 8;4:26. doi: 10.3389/fmed.2017.00026. eCollection 2017. PMID 28337439
- [Background] Voscopoulos CJ, MacNabb CM, Brayanov J, Qin L, Freeman J, Mullen GJ, Ladd D, George E. The evaluation of a non-invasive respiratory volume monitor in surgical patients undergoing elective surgery with general anesthesia. J Clin Monit Comput. 2015 Apr;29(2):223-30. doi: 10.1007/s10877-014-9596-0. Epub 2014 Jul 19. PMID 25037938
- [Background] Bai Y, Xu Z, Chandrashekar M, St Jacques PJ, Liang Y, Jiang Y, Kla K. Comparison of a simplified nasal continuous positive airways pressure device with nasal cannula in obese patients undergoing colonoscopy during deep sedation: A randomised clinical trial. Eur J Anaesthesiol. 2019 Sep;36(9):633-640. doi: 10.1097/EJA.0000000000001052. PMID 31313720